CLINICAL TRIAL: NCT03042026
Title: Developing a Simple Recognition System of Acromegaly
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201204079RIC
Record Dates: First submitted 2017-02-01; First posted 2017-02-03 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-01

CONDITIONS: Acromegaly
MeSH Terms: conditions — Acromegaly

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acromegaly patients: Acromegaly patients
- Healthy subjects: Healthy volunteers

SUMMARY:
We will compare the features of 3D stereophotography of acromegaly patients with that of healthy people. We hope to develop a computerized model to help screening acromegaly patients for early detection and treatment.

DETAILED DESCRIPTION:
Background: Acromegaly is a slowly progressive disease caused by growth hormone (GH) excess. The estimated prevalence of the disease is 40 cases/1000000 population with 3-4 new cases/1000000 population per year. Most patients have classic manifestations due to acral and soft tissue change, including thickening of the calvarium, increased size of frontal sinus, enlargement of the nose, prognathism, and widely spaced teeth. The hands and feet are large, thickened and bulky. Acromegaly was also associated with many comorbidities including cardiovascular complications (acromegalic cardiomyopathy and arterial hypertension), respiratory complications (sleep apnea), metabolic complication (impaired glucose tolerance, diabetes mellitus), joint and bone complications (carpal-tunnel syndrome, osteoarthritis).3 The outcome of growth hormone level suppression after transsphenoidal surgery is far better for microadenomas (80-90%) than for macroadenomas (less than 50%). Furthermore, higher growth hormone level at diagnosis was related to poor prognosis. An early detection of acromegaly with early intervention was desirable. However, due to the slowly progression of the disease, times from symptom onset to diagnosis were 5.2 to 5.9 year4.

Current method to diagnose patients with acromegaly was to check serum GH and insulin-like growth factor 1 (IGF-1). However, tests for growth hormone and IGF-1 are currently unavailable in most hospitals in Taiwan and were expensive. We want to find a better screening tool for acromegaly with less expensive and high efficacy. Due to specific facial appearance of acromegaly, there were studies to recognize acromegaly by computer program1,2,3. They tried to develop computer programs to separate facial photographs of patient with acromegaly and normal subjects. The accuracy could reach 71.9% to 86%. Due to enlarged hand with increased soft tissue in patients with acromegaly, we also want to compare the difference of face, hand and feet morphology and face, hand and feet X ray of acromegaly patients with those of normal population. We hope to set a computer model to early detect acromegaly patients in Chinese people.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-80 years old, Acromegaly patients or Healthy Adults

Exclusion Criteria:

* Pregnancy. Age less than 20 years old or older than 80 years old

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Acromegaly patients and Healthy Adults
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2012-06-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Anthropometry | 1 year from the first time of 3D stereophotography
  Features of the body including face, hands and feet

CONTACTS AND LOCATIONS:
Overall Officials: Shyang-Rong Shih, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No